CLINICAL TRIAL: NCT06661213
Title: Tapinarof for Cutaneous Lupus Erythematosus
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Paras Vakharia, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00222465
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — tapinarof

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tapinarof Treatment (Experimental): CLE participants treated with tapinarof
  Interventions: Drug: Tapinarof

INTERVENTIONS:
Drug: Tapinarof — A thin layer of tapinarof cream is applied to affected areas once daily.
  Other Names: VTAMA

SUMMARY:
The investigators hypothesize that topical application of Tapinarof, an FDA-approved topical Aryl hydrocarbon receptor (AHR) agonist for the treatment of plaque psoriasis, would inhibit lupus-causing T cells and lead to improvement of cutaneous lupus lesions. To test this hypothesis, the investigators will perform a prospective, interventional clinical trial in patients with chronic and/or subacute cutaneous lupus. This trial will include outcomes analyzing the change in cutaneous lupus lesions using standardized assessments, but also analyze pre- and post-treatment skin and blood immune parameters to elucidate the immune effects and changes in lupus as a result of topical AHR agonist application. The goals are to 1) identify if topical AHR agonism leads to improvement in cutaneous lupus, and 2) examine the immunopathology of cutaneous lupus and its alteration with topical AHR agonist treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Patients with a histopathological or clinical diagnosis of chronic and/or subacute CLE
* Patients with at least one active cutaneous lupus lesion with a diameter ≥ 1cm and CLA-IGA-R score of ≥ 3 at screening and baseline

Exclusion Criteria:

* Unwillingness or inability to complete informed consent process or comply with the study protocol
* Patients who are pregnant or breast-feeding
* Other dermatologic diseases whose presence or treatments would interfere with evaluation of the study drug or interpretation of participant safety or trial results
* History of allergy, hypersensitivity reaction, or anaphylaxis to any component of the study drug
* Application to cutaneous lupus lesion(s) being assessed of topical corticosteroids, topical calcineurin inhibitors, or topical janus kinase inhibitors within 1 weeks of study drug initiation
* Application to cutaneous lupus lesion(s) being assessed of topical tapinorof within 4 weeks of study drug initiation
* Prior use of anifrolumab within the last 6 months
* New initiation of systemic immunosuppressive or immunomodulating drugs (e.g. oral or injectable corticosteroids, methotrexate, cyclosporine, mycophenolate mofetil, azathioprine, belimumab), antimalarials (hydroxychloroquine, chloroquine, quinacrine), or systemic janus kinase inhibitors within 12 weeks of study drug initiation
* For patients already on the following treatment(s) prior to enrollment: unstable or changing of dosing of systemic immunosuppressive or immunomodulating drugs (e.g. oral or injectable corticosteroids, methotrexate, cyclosporine, mycophenolate mofetil, azathioprine, belimumab), antimalarials (hydroxychloroquine, chloroquine, quinacrine), or systemic janus kinase inhibitors within 4 weeks of study drug initiation
* Patients with active infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in Cutaneous Lupus Activity (CLA) Investigator Global Assessment (IGA) - Revised (R) score | 16 weeks
  Proportion of participants who achieve 0 or 1 on the CLA-IGA-R scale at Week 16 (5-point Likert scale 0-4, 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe)
Improvement in the CLE Disease Area and Severity Index (CLASI)-Activity (A) score | 16 weeks
  Mean change in CLASI-A from Week 0 to Week 16.The maximum score for CLASI-A is 70 points, with a score of 0-9 indicating mild disease, 10-20 indicating moderate disease, and 21-70 indicating severe disease. A score of 0 indicates no active mucocutaneous lesions

CONTACTS AND LOCATIONS:
Overall Officials: Paras Vakharia, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No